CLINICAL TRIAL: NCT02941471
Title: A Double-blind Pilot Randomised Trial of Transabdominal Interferential Stimulation and Transcutaneous Electrical Nerve Stimulation for Severe Chronic Constipation in Adults Unresponsive to Conservative Treatments
Brief Title: Transabdominal Electrical Stimulation for Constipation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St Mark's Hospital Foundation (Other)
Responsible Party: Principal Investigator, Fareed Iqbal, Clinical Research Fellow/PI, St Mark's Hospital Foundation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: StMarksHF
Record Dates: First submitted 2016-10-18; First posted 2016-10-21 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Constipation
Keywords: Constipation; Neuromodulation; Interferential; Transabdominal
MeSH Terms: conditions — Constipation | interventions — Electric Stimulation Therapy; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interferential Stimulation (Experimental): Medical Device: Interferential stimulation. Stimulation parameters: 4 KHz of carrier stimulation, beat frequency between 80-160Hz, amplitude upto 33mA. Delivered via two 100mm x 50mm adhesive pads placed on the anterior abdominal wall
  Interventions: Device: Interferential Stimulation
- Standard electrical stimulation (Active Comparator): Medical Device: Standard electrical stimulation. Parameters set to provide continuous electrical stimulation at a pulse width of 210µs and a frequency of 14Hz and an amplitude upto 33mA.
  Interventions: Device: TENS stimulation

INTERVENTIONS:
Device: Interferential Stimulation — Transabdominal interferential electrcial stimulation
  Other Names: NeuroTrac® IFC Rehab device (Verity Medical Ltd, UK).
  Arms: Interferential Stimulation
Device: TENS stimulation — Transabdominal standard electrical stimulation
  Other Names: NeuroTrac® Continence device (Verity Medical Ltd, UK).
  Arms: Standard electrical stimulation

SUMMARY:
Several transabdominal electrical stimulation studies have been reported for constipation in childhood. This study aims to assess the efficacy of this technique in adults with chronic constipation and compare two different electrical therapies.

DETAILED DESCRIPTION:
Patients with Rome III defined constipation unresponsive to medical and behavioural treatment will be randomised in a double-blind prospective trial to receive either four weeks of transabdominal electrical stimulation (TENS) or Interferential stimulation (IFC). Treatment will be self-administered at home for sixty minutes a day. The response to treatment will be assessed with the Patient Assessment of Constipation Quality of Life questionnaire (PAC-QOL), the Patient-Assessment of Constipation Symptoms (PAC-SYM) tool and a bowel visual analogue scale (VAS). A bowel diary will be kept a week before and during the final week of stimulation, recording daily bowel frequency.

IFC stimulation is an effective, cheap and low risk intervention which has demonstrated efficacy for dysphagia, urinary incontinence, overactive bladder syndromes and chronic pain. The precise mechanism of its analgesic and pro-kinetic effect is unknown. The intervention is delivered by two separate continuous alternating electrical currents. Two pairs of pad electrodes are arranged in a quadripolar manner where each pair delivers a different frequency of current. It is suggested that this arrangement of stimulation improves colonic propagation. However as direct massage of the abdomen has demonstrated benefit in constipation it is argued that IFC is not a specific requirement and that non-IFC electrical stimulation over the abdomen is sufficient to evoke the same colonic and clinical responses. Owing to these questions the efficacy of this intervention will be further evaluated in adults.

This study has two aims. The primary aim is to evaluate the effectiveness of transabdominal electrical nerve stimulation (TENS) in adult patients with chronic constipation. The secondary aim is to establish whether IFC was superior to non-IFC (TENS) electrical stimulation in adults with chronic constipation.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Rome III defined constipation (frequency of defecation of less than three times a week, straining or sense of incomplete emptying associated with at least 25% of defecations. Lumpy, hard stools or anal digitation for at least 25% of defecations
* Failed Biofeedback
* Competent and willing to complete stimulation at home
* Competent and willing to complete the questionnaires and bowel diaries

Exclusion Criteria:

* Rectal prolapse
* Active inflammatory bowel disease
* Pregnancy or intention to become pregnant during trial
* Spinal cord injuries/cauda equina syndrome
* Other implanted electrical devices
* Allergy to device components
* Neurological disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Patient Assessment of Constipation Quality of Life questionnaire (PAC-QOL) | After 4 weeks of stimulation
  A validated tool for constipation severity assessment

SECONDARY OUTCOMES:
Patient-Assessment of Constipation Symptoms (PAC-SYM) | After 4 weeks of stimulation
  A validated tool for constipation severity assessment
A bowel visual analogue scale | After 4 weeks of stimulation
  a bowel visual analogue scale (0-100 where 0= 'very unhappy' 100= 'very happy') based on patients' response to the question 'how happy are you with the way your bowel has been functioning'
Weekly bowel and laxative diary | one week and 4 weeks of stimulation
  Standard bowel and laxative diary

CONTACTS AND LOCATIONS:
Overall Officials: Alan Warnes, PhD, Study Chair — The London Northwest Healthcare NHS Trust